CLINICAL TRIAL: NCT06508086
Title: LASER ABLATION VERSUS KARYDAKIS TECHNIQUE IN THE TREATMENT OF PILONIDAL SINUS DISEASE: A COMPARATIVE STUDY
Brief Title: Pilonidal Sinus Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Assem Mahmoud Ahmed, Resident, Department of General Surgery, Faculty of Medicine, Sohag University, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-24-06-26MS
Record Dates: First submitted 2024-07-12; First posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Pilonidal Sinus
MeSH Terms: conditions — Pilonidal Sinus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group (A) LASER ABLATION (Active Comparator)
  Interventions: Procedure: laser ablation technique in the treatment of pilonidal sinus
- group (B) KARYDAKIS TECHNIQUE (Active Comparator)
  Interventions: Procedure: Karydakis technique in the treatment of pilonidal sinus

INTERVENTIONS:
Procedure: laser ablation technique in the treatment of pilonidal sinus — group (A) will include patients with pilonidal sinus disease who will be operated by sinus tract ablation procedure using 1470 nm Diode laser
  Arms: group (A) LASER ABLATION
Procedure: Karydakis technique in the treatment of pilonidal sinus — group (B) will include patients with pilonidal sinus disease who will be operated by Karydakis technique
  Arms: group (B) KARYDAKIS TECHNIQUE

SUMMARY:
The aim of this study is to compare the outcomes of Karydakis technique versus sinus tract ablation procedure using 1470 nm Diode laser for the treatment of pilonidal sinus and provide evidence-based guidance to select the most appropriate operative procedure.

ELIGIBILITY:
Inclusion Criteria:

* All patients with a clinical diagnosis of symptomatic uncomplicated pilonidal sinus, males or females, any age will be included in our study.

Exclusion Criteria:

* Patients with pilonidal abscess and any associated acute condition.
* Patients with hidradenitis suppurativa.
* Refusal.
* Unfit for surgery.
* Recurrence.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
recurrence rate in the treatment of pilonidal disease | 6 months after the operation
  the patients undergo follow up at the outpatient clinic for manifestations of recurrence eg. discharge, multiple pits

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

REFERENCES:
- [Background] Guner A, Cekic AB, Boz A, Turkyilmaz S, Kucuktulu U. A proposed staging system for chronic symptomatic pilonidal sinus disease and results in patients treated with stage-based approach. BMC Surg. 2016 Apr 16;16:18. doi: 10.1186/s12893-016-0134-5. PMID 27084534
- [Background] Doll D, Matevossian E, Wietelmann K, Evers T, Kriner M, Petersen S. Family history of pilonidal sinus predisposes to earlier onset of disease and a 50% long-term recurrence rate. Dis Colon Rectum. 2009 Sep;52(9):1610-5. doi: 10.1007/DCR.0b013e3181a87607. PMID 19690490
- [Background] Dessily M, Charara F, Ralea S, Alle JL. Pilonidal sinus destruction with a radial laser probe: technique and first Belgian experience. Acta Chir Belg. 2017 Jun;117(3):164-168. doi: 10.1080/00015458.2016.1272285. Epub 2017 Jan 6. PMID 28056720